CLINICAL TRIAL: NCT00968097
Title: Evaluation of [123I] MNI-340 and SPECT as a Marker of Beta-amyloid Protein Deposition in Subjects With Alzheimer Disease in Comparison to Healthy Subjects
Brief Title: Evaluation of [123I] MNI-340 and SPECT as a Marker of Beta-Amyloid Protein Deposition
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Early Phase I study of [123I]MNI-340 did not evidence as marker of disease
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MNI-340-01
Record Dates: First submitted 2008-04-25; First posted 2009-08-28 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer' disease; SPECT imaging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 123-I MNI-340 — To assess the dynamic uptake and washout of 123-I MNI-340, a potential imaging biomarker for β-amyloid burden in brain

SUMMARY:
The main objectives of this proposal are as follows:

To assess the dynamic uptake and washout of 123-I MNI-340, a potential imaging biomarker for β-amyloid burden in brain, using single photon emission computed tomography (SPECT) in similarly aged Alzheimer's (AD) subjects and healthy controls

To perform blood metabolite characterization of 123-I MNI-340 in healthy and AD subjects to determine the metabolic fate and nature of metabolites in assessment of 123-I MNI-340 as a single photon computed tomography (SPECT) brain imaging agent

DETAILED DESCRIPTION:
Background:

Alzheimer's dementia (AD) is a common disorder of the aging brain causing progressive and irreversible impairment in memory and cognitive function. Beginning with the initial description of Alzheimer's dementia (AD) in 1906 when abnormal accumulations of plaques and tangles in the brain of a woman with severe cognitive impairment were first noted, the pathophysiology of AD has been intimately associated with a progressive neuropathologic process involving abnormal protein deposition in brain. More recent work has implicated the accumulation of β-amyloid as an early feature of AD, which may be directly responsible for some of the clinical manifestations of the disease. Pathologic studies suggest levels of β-amyloid are elevated even in cases classified as having questionable dementia (CDR score = 0.5), and increases in amyloid are strongly correlated with cognitive decline. Increases in β-amyloid precede significant tau pathology suggesting the formation of plaques early in the disease may be of clinical importance.

Until recently post-mortem examination of brain tissues was the only means available for directly evaluating the changes occurring in the brain in AD and related neurodegenerative diseases. In the last decade, the development of highly specific techniques for imaging the brain in AD has expanded our ability to measure the process of the disease over time in a living individual. Briefly, these techniques involve intravenous administration of radioactively-labeled compounds which bind to selective target sites in brain. The scintigraphic imaging methods PET (positron emission tomography) or SPECT (single photon emission computed tomography) are able to detect the spatial distribution of the radioactive compound in the brain and can be used as an objective, sensitive, and accurate method to quantify the concentration of the targets site in different brain regions.

Using these techniques, β-amyloid aggregates have been successfully imaged in several studies in AD patients using high affinity 11-C and 18-F-labeled PET tracers (PIB and FDDNP, AV-1). More recently, another tracer, based on a thioflavin-S derivative, 6-iodo-2-(4'-dimethylamino-)phenyl-imidazol[1,2-a]pyridine, IMPY, labeled with 123-I has been used to image amyloid. MNI-340 has a similar structure to PIB, but the 123-I radioactive tag offers distinct advantages for large-scale clinical imaging studies of β -amyloid plaque targeted treatments as a marker of plaque burden and efficacy of therapeutic intervention. The longer half-life (13.1 h) of 123-I permits imaging in multiple subjects in a single research-dedicated imaging center. This minimizes variability introduced in multicenter quantitative imaging trials where different cameras, image processing methods, and QA procedures all conspire to increase the variance imaging biomarkers. Using this model, our group pioneered a method to evaluate the loss of dopamine function in Parkinson's disease using a radioactive drug 123-I β-CIT, which binds directly to dopamine nerve terminals.

The adaptation of imaging agents like 123-I MNI-340 as a biomarker of β-amyloid deposition in AD patients for assessing disease requires human validation studies. The purpose of this study is to develop and characterize 123-I MNI-340 as an objective biomarker in AD. The significance of this work lies in applying state-of-art quantitative neuroimaging tools to develop a relevant biomarker in living AD patients. In this context we propose to investigate the feasibility of applying this technique as an imaging biomarker of disease in AD patients.

Research Plan:

General Design and Methods. The underlying goal of this study is to assess 123-I MNI-340 SPECT imaging as a tool to detect ß-amyloid deposition in the brain of AD research participants and age- and gender-matched healthy subjects. All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImaging (MNI) in New Haven, CT. Approximately 10 patients with Alzheimers disease (AD) and 10 similarly aged healthy controls will be recruited to participate in this study. Healthy controls will be screened to ensure that there is no evidence of cognitive decline or significant neurological deficit.

Informed consent will be obtained for all subjects. All subjects will undergo a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations. Subjects will be given a bolus injection of 123-I MNI-340 in an antecubital vein. Subjects will undergo serial SPECT imaging scans and serial venous plasma sampling for measurement of 123-I MNI-340 in plasma (both protein bound and free) over a period of up to 8 hours. The quantitative and visual imaging analyses will be performed by an image-processing specialist who will remain blinded to any clinical information.including diagnosis. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, 123-I MNI-340. Time to the peak uptake and amplitude of the peak uptake will be evaluated for all brain regions and the results for the AD patients and controls will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's Subject Selection. Subjects who have a clinical diagnosis of mild to moderate Alzheimer's disease will be recruited for this study. The following criteria will be met for inclusion of AD subjects in this study:

  * The participant is 50 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
  * Mini-Mental Status Exam score > 16 and < 25.
  * Modified Hachinski Ischemia Scale score of ≤ 4.
  * Geriatric Depression Scales (GDS) ≤ 10.
  * For females, non-child bearing potential or negative urine and blood pregnancy test on day of 123-I MNI-340 injection.
* Healthy Control Subject Selection: Healthy control subjects who have no neurological disease will be recruited for this study. The following criteria will be met for inclusion of healthy control subjects in this study:

  * The participant is 50 years or older.
  * Written informed consent is obtained.
  * Negative history of neurological or psychiatric illness based on evaluation by a research physician.
  * Mini-Mental Status Exam score ≥28.
  * For females, non-child bearing potential or negative urine and blood pregnancy test on day of 123-I MNI-340 injection.

Exclusion Criteria:

* Alzheimer's subjects will be excluded from participation for the following reasons:

  * The subject has signs or symptoms of another neurodegenerative disease including Parkinson's disease, diffuse Lewy body dementia, or history of significant cerebrovascular disease.
  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
  * The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * The subject has participated in another clinical study within the previous 30 days.
  * Clinically significant MRI evidence of vascular disease or alternative neurologic disorder
  * Pregnancy
* Healthy control subjects will be excluded from participation for the following reasons:

  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
  * The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * The subject has participated in another clinical study within the previous 30 days.
  * Pregnancy
  * Clinically significant MRI evidence of vascular disease or neurologic disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, 123-I MNI-340. | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Danna L Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- The Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States